CLINICAL TRIAL: NCT01300988
Title: A Phase Ib, Randomized, Placebo Controlled, Double Blind Study to Determine the Safety, Viral Suppression, Pharmacokinetics and Immune Modulatory Effects of Treatment With Aprepitant (Emend®) in HIV Infected Individuals
Brief Title: Effects of Treatment With Aprepitant (Emend®) in HIV Infected Individuals. 375 mg Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 811938; U01MH090325 (NIH)
Record Dates: First submitted 2010-12-16; First posted 2011-02-23 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: HIV Infection
Keywords: HIV infection; Neurokinin-1 receptor antagonist; CCR5 expression; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aprepitant (Active Comparator): Aprepitant (Emend®) 375 mg daily for 14 days
  Interventions: Drug: Aprepitant
- Placebo (Placebo Comparator): Aprepitant (Emend®) placebo for 14 days
  Interventions: Drug: Aprepitant placebo

INTERVENTIONS:
Drug: Aprepitant — Aprepitant (Emend®) 375 mg daily for 14 days
  Arms: Aprepitant
Drug: Aprepitant placebo — Aprepitant(Emend®) placebo for 14 days
  Arms: Placebo

SUMMARY:
The investigators' in vitro data suggest that Neurokinin-1 receptor antagonists like aprepitant will decrease the expression of CCR5, an essential co-receptor in the life cycle of HIV, in the surface of macrophages and lymphocytes to levels at least similar to those observed in patients heterozygous for the CCR5 32 mutation. Together with a direct potential antiviral effect this could alter disease progression in patients with HIV infection.

The investigators' hypothesis is that aprepitant is safe, tolerable and has antiviral activity in HIV infected individuals.

This is randomized, placebo controlled, double blind study to determine the safety and antiviral activity of aprepitant by comparing the change in HIV RNA viral load after 2 weeks of aprepitant monotherapy.

18 HIV infected males and females ≥ 18 years old who have early infection with CD4 cell counts ≥ 350 cells/mm3. Subjects will be randomized 1:1 to receive 375 mg of aprepitant (Emend®) or placebo.

DETAILED DESCRIPTION:
DESIGN

Randomized, placebo controlled, double blind study to determine the safety and antiviral activity of aprepitant by comparing the change in HIV RNA viral load after 2 weeks of aprepitant monotherapy.

DURATION

42 days.

SAMPLE SIZE and POPULATION

18 HIV infected males and females ≥ 18 years old who have early infection with CD4 cell counts ≥ 350 cells/mm3.

REGIMEN

Subjects will be randomized 1:1 to receive aprepitant (Emend®) or placebo.

Arm A: Aprepitant placebo Arm B: Aprepitant 375 mg QD

HYPOTHESIS AND STUDY OBJECTIVES

Hypothesis : Aprepitant is safe, tolerable, and has antiviral activity in HIV infected individuals.

Primary Objectives:

To assess the safety and tolerability of 375 mg aprepitant for 2 weeks To assess the response of plasma HIV-1 RNA to 375 mg of aprepitant compared with baseline.

Secondary Objectives:

To investigate the course and duration of antiretroviral response 375 mg of aprepitant given over a 14-day period.

To evaluate the dose-response and pharmacokinetic and pharmacodynamic relationship between viral RNA change and aprepitant plasma levels.

To evaluate aprepitant effects on CD4+ and CD8+ T-cell counts, circulating SP levels, natural killer cell number and function and CCR5 expression in peripheral PBMCs.

To evaluate the effects of aprepitant in the viral tropism and envelope sequence of the main HIV-1 population of the participants.

To assess viral drug susceptibility in conjunction with baseline coreceptor tropism phenotype and changes in coreceptor phenotype after the exposure to aprepitant.

To evaluate aprepitant effects on fasting plasma glucose, insulin, HDL, free fatty acids, and triglyceride concentrations after 14 days of treatment.

To provide preliminary description of any change from baseline in sleep quality, anxious mood, depressed mood and neurocognitive measures after 2 weeks of aprepitant therapy.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, as documented by a rapid HIV test or any FDA-Approved HIV-1 Enzyme or Chemiluminescence Immunoassay (E/CIA) test kit and confirmed by Western blot at any time prior to study entry.
* CD4+ cell count >= 350/mm3 obtained within 90 days prior to study entry
* Plasma HIV-1 RNA of >=2,000 copies/mL as measured by any standard assay and performed within 90 days prior to study entry.
* CCR5 tropic virus exclusively as determined by the Monogram tropism assay (PhenoSense Entry™) to be performed within 90 days of study entry.
* Laboratory values obtained within 30 days prior to study entry, as follows:

  * Absolute neutrophil count (ANC) >= 750/mm3
  * Hemoglobin >= 10.0 g/dL
  * Platelet count >= 100,000/mm3
  * Creatinine <= 2 x ULN
  * AST (SGOT), ALT (SGPT), and alkaline phosphatase <= 2 x ULN
  * Total bilirubin <= 2.5 x ULN
  * Albumin >= 3 g/dL
* Female subjects of reproductive potential must have a negative spot urine pregnancy test result (with a sensitivity of at least 50 mIU/mL) performed at entry, prior to starting initial study treatment.
* All subjects must agree not to participate in a conception process while on study drug and for 30 days after stopping the medication.
* Karnofsky performance score >= 80 within 30 days prior to study entry.
* Men and women > 18 years of age.
* Ability and willingness of subject to give written informed consent.
* Willing to return for a follow-up visit on day 42.
* Subjects taking any precautionary concomitant medications must be on stable doses for >8 weeks prior to study entry and have no plans to change medications or doses for the duration of the study.

Exclusion Criteria:

* Receipt of antiretroviral treatment within the 16 weeks prior to study entry or intent to initiate antiretroviral therapy within 60 days after entry.
* Diabetes requiring treatment with oral hypoglycemics or insulin therapy.
* Pregnancy within 90 days prior to study entry.
* Breast-feeding.
* Use of drugs that are inhibitors or inducers of metabolism by the cytochrome P450 CYP3A4 or CYP2C9 (such as warfarin and phenytoin) within 7 days of study entry.
* Use of systemic corticosteroids or hormonal agents within 90 days prior to study entry.
* Use of any immunomodulator, HIV vaccines, or investigational therapy within 90 days prior to study entry.
* Any vaccination within 30 days prior to study entry.
* Use of systemic cytotoxic chemotherapy within 90 days prior to study entry.
* History of allergy to aprepitant or its formulations.
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* History of chronic active hepatitis B or C infection or severe hepatic dysfunction (Child-Pugh score > 9) regardless of etiology
* Serious illness requiring systemic treatment and/or hospitalization until subject either completes therapy or is clinically stable on therapy, in the opinion of the investigator, for at least 14 days prior to study entry.
* Weight < 40 kg or 88 lbs. within 90 days prior to study entry.
* History of severe psychiatric comorbidities, such as depression, schizophrenia, mania, psychosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Virologic: Change in log10 HIV-1 RNA from baseline to Day 14 | 14 days
  For the purposes of assessing the primary analysis of efficacy of aprepitant in reducing viral load we will be assessing the difference between the log10 viral load at baseline and at 4 weeks, and constructing a 95% confidence interval around this mean difference within each dose group.
Safety: Incidence of Grade 2, 3, and 4 adverse events | 42 days
  The frequency of grade 2,3 and 4 adverse events for the duration of the study will be measured to assess the safety of the compund in this population. Exact binomial confidence intervals will be calculated around the event rates for any individual adverse events that occur and for the overall rate of adverse events within each body system. For each patient the highest grade occurring adverse event within each body system will be assessed. Tables for adverse events by body system and severity of adverse event will be constructed.

SECONDARY OUTCOMES:
Pharmacokinetic | 14 days
  Individual patient data will be summarized using a noncompartmental analysis (NCA) approach as well as a model-based approach.
Immunologic | 14 days
  A descriptive analysis of the following parameters by arm at each time point will be done:
  * CCR5 mRNA copy number per cell and CCR5 density by flow cytometry.
  * CD4+ cell count at baseline, Days 3, 7, 10, 14, and 42.
  * Time to permanent discontinuation of study treatment for any reason.
  * Baseline coreceptor phenotype (CCR5, CXCR4, or mixed).
  * Time to change from CCR5-only virus to mixed CCR5/CXCR4 or CXCR4-only virus as detected by the phenotype/genotype assays that will be used in this study.
Neurologic | 14 days
  Evaluate individual changes from baseline to 14 days for these subjects in the HAM-D 17 Depression Rating Scale score, the HAM-A, and the PSQI

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Tebas, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Clinical Trials Unit. University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Lai JP, Ho WZ, Zhan GX, Yi Y, Collman RG, Douglas SD. Substance P antagonist (CP-96,345) inhibits HIV-1 replication in human mononuclear phagocytes. Proc Natl Acad Sci U S A. 2001 Mar 27;98(7):3970-5. doi: 10.1073/pnas.071052298. PMID 11274418
- [Background] Lai JP, Ho WZ, Kilpatrick LE, Wang X, Tuluc F, Korchak HM, Douglas SD. Full-length and truncated neurokinin-1 receptor expression and function during monocyte/macrophage differentiation. Proc Natl Acad Sci U S A. 2006 May 16;103(20):7771-6. doi: 10.1073/pnas.0602563103. Epub 2006 May 4. PMID 16675550
- [Background] Ho WZ, Evans DL, Douglas SD. Substance P and Human Immunodeficiency Virus Infection: Psychoneuroimmunology. CNS Spectr. 2002 Dec;7(12):867-874. doi: 10.1017/s1092852900022483. PMID 12766696
- [Background] Ho WZ, Lai JP, Li Y, Douglas SD. HIV enhances substance P expression in human immune cells. FASEB J. 2002 Apr;16(6):616-8. doi: 10.1096/fj.01-0655fje. PMID 11919172
- [Background] Li Y, Douglas SD, Song L, Sun S, Ho WZ. Substance P enhances HIV-1 replication in latently infected human immune cells. J Neuroimmunol. 2001 Dec 3;121(1-2):67-75. doi: 10.1016/s0165-5728(01)00439-8. PMID 11730941